CLINICAL TRIAL: NCT04653259
Title: Using the LyfeMD Application for Effective Maintenance of Remission and Improved Quality of Life in Crohn's Disease and Ulcerative Colitis: A Randomized Controlled Trial
Brief Title: Digital Nutrition Therapy for Patients With IBD
Acronym: LYFEMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Maitreyi Raman, Clinical Associate Professor, Director Clinician Investigator Program (CIP), Medical Director Alberta's Collaboration of Excellence for Nutrition in Digestive Diseases (Ascend) , Medical Director Nutrition Services, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB20-1534
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The INT group will meet with their health coach over the phone or video chat. The health coach will orient them to the LyfeMD, app and ensure the participant has received a nutrition plan in the app. They will be asked to complete the app assessment tools to design a personalized nutrition, physical activity and yoga and meditation program. They will set goals in each area they are interested in implementing. The health coach will then follow-up by phone, video or email 2 weeks after the initial meeting, then monthly with the patient for 2 more months (total of 4 meetings). The health coach will use the following schedule to discuss app related content: First visit nutrition content; second visit behaviour change tools; third visit Yoga, meditation and breathing plans, and; the fourth visit the physical activity plans. The health coach will also be available to answer questions when required using email. Goal attainment will be collected weekly within the app.
  Interventions: Other: LYFE MD app
- Conventional Management Group (No Intervention): The CM group (n=22) will receive conventional care as well as a similar health coaching schedule as the intervention group. The health coach will meet the patient over the phone or video chat to outline their role over the next 3 months and to provide general nutrition guidelines using Canada's Food Guide and Alberta Health Services online resources. The health coach will then follow-up by phone, video chat or email 2 weeks after the initial meeting, then monthly with the patient for 2 more months (total of 4 meetings). The health coach session topics will be the same as the intervention group. For example, the second visit will provide online resources from Alberta Health Services focused on promoting behaviour change, the third visit will orient the patient to Alberta Health Services focused online stress management tools and the final visit will share online versions of the Canadian guidelines for physical activity and sedentary time.

INTERVENTIONS:
Other: LYFE MD app — LyfeMD app is a digital health platform for patients living with both Crohn's disease (CD) and Ulcerative colitis (UC). LyfeMD is meant to help people live and thrive while managing their inflammatory disease with holistic, easy-to-implement, evidence based lifestyle therapies. LyfeMD is one app with multiple features - ranging from customized diet using anti-inflammatory principles identified from recent research, exercise plans to mindfulness and stress reduction programs. It helps patients make therapeutic diet choices to treat inflammation and provides stress reduction strategies when they feel unwell. The LyfeMD app also supports patients to maintain remission even when they're feeling well with trusted resources designed to keep them symptom free.
  In addition to delivering personalized and interactive support, the app uses behaviour science to help patients change their habits, improve their health and reduce the burden IBD places on their lives.
  Arms: Intervention Group

SUMMARY:
Background: Alberta's Center of Excellence for Nutrition in Digestive Diseases (Ascend) is dedicated to generating new discoveries regarding the link between nutrition and digestive diseases and mobilizing existing research to change the way physicians treat conditions such as inflammatory bowel disease, cirrhosis and intestinal failure. Ascend is a collaboration of excellence within the Department of Medicine, Division of Gastroenterology at both the University of Calgary and University of Alberta. Dr. Raman, PI, is the Director of Ascend.

One of Ascend's primary initiatives is the development of a digital health platform for patients living with both Crohn's disease (CD) and Ulcerative colitis (UC). Dr. Raman and her team have developed an app called LyfeMD, by translating leading scientific research into a practical and engaging digital format. LyfeMD is meant to help people live and thrive while managing their inflammatory disease with holistic, easy-to-implement, evidence based lifestyle therapies. LyfeMD is one app with multiple features - ranging from customized diet using anti-inflammatory principles identified from recent research led by Dr. Raman's team, and exercise plans to mindfulness and stress reduction programs. It helps patients make therapeutic diet choices to treat inflammation and provides stress reduction strategies when they feel unwell. The LyfeMD app also supports patients to maintain remission even when they're feeling well with trusted resources designed to keep them symptom free.

In addition to delivering personalized and interactive support, the app uses behavior science to help patients change their habits, improve their health and reduce the burden IBD places on their lives. With proprietary research and a team made up of internationally recognized leaders in the gastrointestinal field, LyfeMD is poised to be the trusted digital health solution for people living with IBD.

DETAILED DESCRIPTION:
Study Objectives:

1. To identify if the LyfeMD app improves diet quality, perceived stress, depression, anxiety, well-being, quality of life, sleep, and physical activity minutes.
2. To identify if the LyfeMD app helps improve intestinal inflammation measured by fecal calprotectin in CD and UC patients in clinical remission.

Methods:

This 1-year study at the University of Calgary (n=44) will have a RCT study design. Participants will be randomly allocated to receive the intervention LyfeMD mobile application (INT) for 12-weeks or conventional management (CM) from the IBD clinic at the Foothills hospital.

Intervention Group(INT): The INT group (n=22) will meet with the health coach over the phone or video chat. The health coach will orient the participant to the LyfeMD app, answer technology related questions and ensure that the participant has received a nutrition plan in the app. Participants will be asked to complete the app assessment tools to design a personalized nutrition, physical activity and yoga and meditation program. Participants will set goals in each area that they are interested in implementing.

The health coach will then follow-up by phone, video chat or email 2 weeks after the initial meeting, then monthly with the participants for 2 more months (total of 4 meetings). The health coach will use the following schedule to discuss app related content: First visit nutrition content; second visit behaviour change tools; third visit Yoga, meditation and breathing plans, and; the fourth visit the physical activity plans. The health coach will also be available to answer questions when required using email. Goal attainment will be collected weekly within the app.

Conventional Management (CM): The CM group (n=22) will receive conventional care as well as a similar health coaching schedule as the intervention group. The health coach will meet the patrticipants over the phone or video chat to outline their role over the next 3 months and to provide general nutrition guidelines using Canada's Food Guide and Alberta Health Services online resources. The health coach will then follow-up participant by phone, video chat or email 2 weeks after the initial meeting, then monthly for 2 more months (total of 4 meetings). The health coach session topics will be same as the intervention group. For example, the second visit will provide online resources from Alberta Health Services focused on promoting behaviour change, the third visit will orient the patient to Alberta Health Services focused online stress management tools and the final visit will share online versions of the Canadian guidelines for physical activity and sedentary time.

The health coach will be available to answer questions when required using email.

Following completion of the 12-week study, participants in the control group will receive complimentary access to the LyfeMD app for 12-weeks.

Both groups will meet with the study coordinator face to face at the start and end of the study (13th week). At this time, participants will be given all the study materials they need.

Relationship to Pfizer:

From a Pfizer perspective, the investigators recognize that Inflectra is growing in market share. The LyfeMD program will be used together, in a complementary way alongside biologic therapy. The recent diet study led by the principle investigator indicates that the customized diet using anti-inflammatory principles will induce remission in 6 weeks and maintain remission in patients with CD. The investigators would expect that combining diet therapy with biologics would bolster the effect of the biologic and longevity of remission. With the wellness additions (physical activity and yoga/meditation programs), the investigators predict patients will lead happier lives.

Investigators believe that the LyfeMD app will fill a current gap in the market. The availability of Registered Dietitian (RD), Exercise Physiologists, and Certified yoga and meditation instructors in AB/Canada is inadequate to provide care to every patient with IBD in a convenient and personalized way.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients with ileal, ileo-colonic, or colonic luminal CD and UC in clinical remission (Harvey Bradshaw Index <5 or Partial Mayo Score <3) will be invited to participate.
* Ability to provide informed consent
* Have smart phones to use the app

Exclusion Criteria:

* Patients more than 80 years old.
* Patients will be excluded if they are known to have upper GI Crohn's disease, fistulizing phenotype, > 1 small bowel resection, colectomy, or any psychiatric or neurocognitive comorbidity that would limit compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Short-form 12-items (SF-12): Change is being assessed. | Baseline and 12 week
  Assess quality of life
Perceived stress score 10-item measure (PSS-10): Change is being assessed. | Baseline and 12 week
  measure the stress level
Pittsburgh sleep quality index a validated 10-item sleep score (PSQI): Change is being assessed. | Baseline and 12 week
  Measure the sleep quality
Godin, a validated 4-item tool: Change is being assessed. | Baseline and 12 week
  Physical activity minutes will be measured, to estimate weekly physical activity minutes from both moderate and vigorous leisure-time activity.
24-item tool from the National Institute for Neurological Disorders and Stroke: Change is being assessed. | Baseline and 12 week
  To measure the well being and positive aspect
Generalized anxiety disorder 7-item (GAD-7) tool: Change is being assessed. | Baseline and 12 week
  To measure the anxiety severity
Patient health questionnaire 9-item (PHQ-9) tool: Change is being assessed. | Baseline and 12 week
  To measure depression
Behaviour compliance: Change is being assessed. | Once every week starting from date of randomization upto week 12
  This will be measured by scoring how many goals the patients reports successfully tracking each week in the three different content areas. This is all done inside of the app.

SECONDARY OUTCOMES:
24 hour ASA food recalls: Change is being assessed. | Base line and 12 week
  Assess diet quality
Fecal calprotectin: Change is being assessed. | Baseline and 12 week
  FCP is a test used to detect inflammation in the colon and is associated with disease activity and severity.
Harvey Bradshaw Index (HBI) fro Crohn's disease: Change is being assessed. | Baseline and 12 week
  HBI is a validated, non-invasive measure of disease activity captured through a symptom questionnaire and is a surrogate to endoscopic assessment to determine disease severity. HBI minimum value is "0" and maximum no limit. HBI < 5 is used in this study to indicate clinical remission. HBI> 16 means severe disease activity. Higher scores means worse outcomes. Based on experience with past recruitment for clinical trials, endoscopic assessment is not feasible due to access and patient acceptance.
Partial-Mayo score for ulcerative colitis: Change is being assessed. | Baseline and 12 week
  Partial Mayo Score (PMS), is a bedside measure of disease activity captured through a symptom questionnaire. It uses the three non-invasive components of the full Mayo Score (stool frequency, rectal bleeding and Physician's global assessment). This excludes the score for the endoscopic findings, therefore the maximum score is reduced from 12 to 9 points (1,2).

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Raman, MD, Principal Investigator — University of Calgary
Locations (1):
- TRW building, Foothills, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers outside of the study team.